CLINICAL TRIAL: NCT04336553
Title: Social Prescribing in Sweden (SPiS)- An Interventional Research Project Evaluating a Swedish Model
Brief Title: Social Prescribing in Sweden (SPiS)
Acronym: SPiS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: Forte (Industry)
Responsible Party: Principal Investigator, Ingeborg Nilsson, Professor, Umeå University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1:1
Record Dates: First submitted 2020-04-02; First posted 2020-04-07 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Loneliness
Keywords: Loneliness; Older adults; Social occupations; Participation; Social prescribing

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Social prescribing in sweden (SPiS) (Experimental): Patients (older adults experiencing loneliness) at a Health care clinic are invited to an optional additional internal referral for social prescribing (SPiS) within four working days. SPiS is a means of enabling the professionals to refer people to a range of local, non-clinical services. SPiS will involve a variety of activities, tailored to the patients needs and desires) which are typically provided by voluntary and community sector organisations.
  Interventions: Behavioral: Social prescribing in Sweden (SPiS)
- Control: Social prescribing in sweden (SPiS) (No Intervention): Patients (older adults experiencing loneliness) at a Health care clinic are invited to an optional additional internal referral for social prescribing (SPiS) within three months. SPiS is a means of enabling the professionals to refer people to a range of local, non-clinical services. SPiS will involve a variety of activities, tailored to the patients needs and desires) which are typically provided by voluntary and community sector organisations.

INTERVENTIONS:
Behavioral: Social prescribing in Sweden (SPiS) — Social prescribing in sweden (SPiS)
  Arms: Intervention: Social prescribing in sweden (SPiS)

SUMMARY:
Loneliness among older adults has become an issue of public concern, as it is associated with increased morbidity and mortality. Yet, despite the urgency, there is little information on how to reduce or prevent loneliness. The focus of this project is using experiences from the United Kingdom's initiative social prescribing, which gives General Practitioners the option of referring clients in need to a coordinator, who in dialogue with the client finds activities for the client to engage in within the local community. Until now, social prescribing has not been tested in Sweden. Therefore, with the overarching goal of reducing loneliness and improving health and wellbeing, the aim of the project is to develop and test a Swedish social prescribing program in order to explore circumstances under which the program can reduce loneliness and improve wellbeing in older adults. The project will be carried out in collaboration between researchers, a primary healthcare center, and a community activity initiative. In the first phase, the research group will bring potential end-users and stakeholders together in workshops to discuss, develop, and design a Swedish program for social prescribing. Interviews with potential end-users and stakeholders will be carried out to analyze challenges and possibilities with the program. In a second phase, the Swedish program will be implemented to evaluate experiences and the effect of Social prescribing in Sweden regarding loneliness, health, wellbeing among older adults (65 yrs or older) in Sweden. The study will be carried out in a feasibility study and a large-scale RCT study. including both qualitative and quantitative data Based on the results of this study, there will be new knowledge gained concerning if and how social prescribing can be used among older adults in a Swedish context.

DETAILED DESCRIPTION:
Loneliness among older adults has become an issue of public concern. There seems to be a high and stable prevalence of reported loneliness, with as many as 50% of older adults reporting serious or moderate loneliness. There is also growing evidence on the significant harmful effects of loneliness in older adults . Although the situation is urgent, no specific type of intervention has demonstrated a robust evidence base for reducing loneliness. There are, however, promising initiatives that manage to take the wider context in which the individual lives into account. Initiatives such as Social Prescribing in the United Kingdom identify the individual's needs, and guide them in getting involved with their community, by linking people with local supportive social activities and opportunities. However, such initiatives are sensitive to context, and may not be easily transferred between national contexts. The focus of this project is to develop and implement Social Prescribing in a Swedish context, as this has not yet been done. Our novel contribution to this field is: a) developing a Swedish version of a social prescribing method together with potential end-users and stakeholders; and b) evaluating the first test and implementation of this method. Thus, this project has the potential to develop important knowledge regarding how to prevent and/or reduce an urgent public health issue, loneliness among older adults, in a non-medical way via social prescribing in a Swedish context.

Background and point of departure

Systematic reviews show that social isolation and loneliness among older people is a substantial problem (affecting 7-17% and 40% respectively), and that lack of social inclusion and a feeling of loneliness negatively affects physical and mental health. These issues are especially prevalent in older people with health problems, and are associated with socio-demographic factors (gender) and social factors (e.g., civil status and meaningful social contacts). The research findings call for attention to be given to the provision of services for meeting societal ideals in caring for the older generation, confronting the rising isolation and subjective loneliness which harms individual health and burdens national and global economies.

There might though be protective factors addressing loneliness as research demonstrates the importance of social relations and social engagement in older people's health, well-being, and cognitive health. Strong mortality effects also exist,148 longitudinal studies revealed a 50% mortality reduction in persons with strong social relationships.

Societal services need to be developed that prevent loneliness and support social participation. A social equivalent to the physical activity on prescription is the United Kingdom initiative started in 2002 called social prescribing, which serves as a way of linking patients in primary care with sources of support within their local community. Social prescribing concerns expanding the options available to General Practitioners (GP) by allowing them to forward a client with psychosocial issues to existing meaningful activities in the community that meet these needs. There are no set standards in the procedures of social prescribing, but it gives a GP the option of using a non-medical referral, either as a stand-alone, or together with existing treatments. The sources of support in the community can be either in the volunteer or community sectors. Challenges that have been described include the multiplicity of options and the logistical difficulties although the idea is simple, the implementation is complex. What is essential is that there is a direct referral from primary care, and an identified coordinator who connects the person to local activities that meet their needs and aspirations.

Although no robust evidence, findings report that social prescribing is broadly supportive to reducing demand on primary and secondary care, and has the potential to deliver cost savings, improvements in wellbeing, reduction of mental and physical symptoms, as well as a reduction in social isolation and loneliness. There is, in particular, a need to highlight research questions such as; When, for whom, and how well does social prescribing work, and in addition, what effect does it have?

Social prescribing has not yet been tested in a Swedish context. There are reasons to believe that perceptions will differ somewhat between the two countries, partly as a consequence of their different ways of understanding relations between the citizen and the "proper" provider of healthcare. With a high number of older adults reporting loneliness, and knowing the harmful effects of this situation, initiatives need to be taken. Social prescribing developed and implemented into a Swedish context is such an initiative.

In the first phase, the researchers will develop and design a social prescribing intervention for a Swedish context (SPiS) and in the second phase, the theory will then be tested while the intervention is implemented in a regular primary healthcare center to assess how the program works. Finally, in a third phase, the program theory will be refined based on the prior developed knowledge.

Co-creation together with a feasibility study and a randomized controlled trial will be used in order to understand and reflect design and development of program for social prescribing.

Both quantitative as well as qualitative data will be collected using different methods. In order to understand feasibility and reach power in the statistics, the program will be implemented in at least eight different primary care centers around Sweden. Randomly older adults will be selected to either get Social prescribing within four working days (intervention group) or be on a waiting list (control group) for three months.

Individual interviews

Group interviews will be performed with representatives from our collaborating partners; a) the health care center, b) the involved community-based activity initiative, and c) local and societal representatives for older adults (65 years old or older) in order to gain knowledge about factors important to address loneliness, health and well-being. Questions about the theoretical underpinnings of the model, the practical implementation of the model in the regular day to day practice as well as the fidelity to the prescription will be important topics to address. Social prescribing per se and its potential effective mechanisms, moderating factors, as well as barriers in the procedure will also be discussed with the profession and stakeholders.

In addition, qualitative interviews will be conducted with the participants who have received social prescribing as well as the professionals who deliver the intervention.

Quantitative measures

Quantitative demographic data of the participants (older adults receiving the SPiS), age, gender, education level, diagnosis affecting activity performance and interests, will be collected at baseline and follow-up followed by measurement of loneliness, self-rated health, mapping of social networks and social support.

Data analysis

The quantitative data will generate evidence regarding the expected outcomes of loneliness, health and activity engagement to address the issue of for whom, under which circumstances, and in what respect the intervention is working. Descriptive statistics, as well as parametric and non-parametric statistical analysis will be used to detect changes between groups of older adults in the outcome variables.

Evidence generated through the qualitative work focusing particularly on contextual factors and potential mechanisms will address the issue of what in the intervention is working and why. Data will be analyzed thematically, with grounded theory approaches and/or other relevant qualitative measures.

ELIGIBILITY:
Inclusion Criteria:

- Persons 65 years or older who experience loneliness will be included after given informed consent

Exclusion Criteria:

- Persons who, due to cognitive impairment, are unable to give informed consent will be excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Loneliness | 0, 3 and 12 month
  The UCLA loneliness scale used for studying changes in loneliness interventions, using this scale, participants' self-reported experiences of loneliness will be measured. The measurement includes 20 statements, rated on a four-step scale from never to always. The given scores are summarized into a total score, ranging from 20-80. Four levels of loneliness have been identified and preliminarily established, and the measurement has been used on groups of older people, and frequently in intervention studies.

SECONDARY OUTCOMES:
Health | 0, 3 and 12 months
  Change in Self-rated general health will be assessed using the visual analogue scale (VAS) from the EQ-5D scale. The VAS is a psychometric response scale which measures subjective characteristics or experiences in a qualitative way. When responding to the VAS item in this project, the respondents specify their level of agreement to the statement "in general how do you experience your health?" by indicating a position along a continuous line between the two end-points, "best possible health and worst possible health".
Health | 0, 3 and 12 months
  Short Form Health Survey Swedish version (SF-12), will be used to capture the overall change of subjective health status. The SF-12 is a questionnaire covering physical health and mental well-being. SF-12, developed from SF-36, has established validity and reliability for use in older populations, and has a similar responsiveness to change as SF-36
Depression | 0, 3 and 12 months
  The GDS-15, depression scale is used to identify changes in symptoms of depression in older adults. The GDS consists of 15 self-rated questions that will assess the level of enjoyment, interest social interaction and more among the older adults. In order to screen for symptoms of depression rather than factors associated with aging, the GDS focuses specifically on psychiatric rather than somatic symptoms.
MNPS Interest checklist | 0, 3 and 12 months
  The checklist is used to identify changes in leisure engagement. The MNPS interest checklist consist of 20 self-rated questions of interest, doing, motivation and well-being from pre-set leisure activities
Social network and support | 0, 3 and 12 months
  Questions related self-rated experiences of social network and support from social network

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Nilsson, Principal Investigator — Umeå University
Locations (1):
- Hälsocentralen Husläkarna, Umeå, Sweden

REFERENCES:
- [Background] Nyqvist F, Cattan M, Conradsson M, Nasman M, Gustafsson Y. Prevalence of loneliness over ten years among the oldest old. Scand J Public Health. 2017 Jun;45(4):411-418. doi: 10.1177/1403494817697511. Epub 2017 Apr 6. PMID 28381194
- [Background] Holt-Lunstad J, Smith TB, Baker M, Harris T, Stephenson D. Loneliness and social isolation as risk factors for mortality: a meta-analytic review. Perspect Psychol Sci. 2015 Mar;10(2):227-37. doi: 10.1177/1745691614568352. PMID 25910392
- [Background] Holt-Lunstad J, Smith TB, Layton JB. Social relationships and mortality risk: a meta-analytic review. PLoS Med. 2010 Jul 27;7(7):e1000316. doi: 10.1371/journal.pmed.1000316. PMID 20668659
- [Background] Mann F, Bone JK, Lloyd-Evans B, Frerichs J, Pinfold V, Ma R, Wang J, Johnson S. A life less lonely: the state of the art in interventions to reduce loneliness in people with mental health problems. Soc Psychiatry Psychiatr Epidemiol. 2017 Jun;52(6):627-638. doi: 10.1007/s00127-017-1392-y. Epub 2017 May 20. PMID 28528389
- [Background] Masi CM, Chen HY, Hawkley LC, Cacioppo JT. A meta-analysis of interventions to reduce loneliness. Pers Soc Psychol Rev. 2011 Aug;15(3):219-66. doi: 10.1177/1088868310377394. Epub 2010 Aug 17. PMID 20716644
- [Background] Social prescribing: community-based referral in public health. Perspect Public Health. 2018 Jan;138(1):18-19. doi: 10.1177/1757913917736661. No abstract available. PMID 29290159
- [Background] Dickens AP, Richards SH, Greaves CJ, Campbell JL. Interventions targeting social isolation in older people: a systematic review. BMC Public Health. 2011 Aug 15;11:647. doi: 10.1186/1471-2458-11-647. PMID 21843337
- [Background] Dahlberg L, Andersson L, McKee KJ, Lennartsson C. Predictors of loneliness among older women and men in Sweden: A national longitudinal study. Aging Ment Health. 2015;19(5):409-17. doi: 10.1080/13607863.2014.944091. Epub 2014 Aug 15. PMID 25126996
- [Background] World Health Organization. Knowledge translation on ageing & health: A framework policy development 2012. Geneva, Switzerland.: WHO Document Production Services 2012.
- [Background] Ferlander S. The importance of different forms of social capital for health. Acta Sociologica. 2007;50(2):115-28.
- [Background] Thomson LJ, Camic PM, Chatterjee HJ. Social prescribing: A review of community referral schemes. London: University College London: University College London; 2015
- [Background] Brandling J, House W. Social prescribing in general practice: adding meaning to medicine. Br J Gen Pract. 2009 Jun;59(563):454-6. doi: 10.3399/bjgp09X421085. No abstract available. PMID 19520038
- [Background] Bickerdike L, Booth A, Wilson PM, Farley K, Wright K. Social prescribing: less rhetoric and more reality. A systematic review of the evidence. BMJ Open. 2017 Apr 7;7(4):e013384. doi: 10.1136/bmjopen-2016-013384. PMID 28389486
- [Background] Wilson P, Booth A. Evidence to inform the commissioning of social presribing. York: University of York. Center of Reviews and Dissemination; 2015.
- [Background] Kimberlee RH. Developing a social prescribing approach for Bristol. Bristol: University of the West of England; 2013.
- [Background] Polley M, Bertotti B, Kimberlee R, Pilkington K, Refsum C. A review of the evidence assessing impact of social prescribing on healthcare demand and cost implications. University of Westminister; 2017.
- [Background] Lindberg J, Lundgren A-S. Positioning the ageing subject: Articulations of choice in Sweden and UK health and social care. Policy studies. 2019:doi.org/10.1080/01442872.2019.1599839.
- [Background] Nilsson I, Nyqvist F, Gustafson Y, Nygard M. Leisure Engagement: Medical Conditions, Mobility Difficulties, and Activity Limitations-A Later Life Perspective. J Aging Res. 2015;2015:610154. doi: 10.1155/2015/610154. Epub 2015 Aug 5. PMID 26346706